CLINICAL TRIAL: NCT04243330
Title: Examining the Effectiveness of an Adaptive Implementation Intervention to Improve Uptake of the VA Suicide Risk Identification Strategy (PEC 19-303)
Brief Title: Adaptive Implementation Intervention for VA Suicide Risk Identification Strategy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: PEX 19-005; PEC 19-303 (Other Grant/Funding Number: VA Quality Enhancement Research Initiative (QUERI))
Record Dates: First submitted 2020-01-10; First posted 2020-01-28 (Actual); Results first posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Suicide
Keywords: prevention; implementation science
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Intervention Model Description: Sequential Multiple Assignment Randomized Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Implementation as Usual (No Intervention): Implementation support consisting of clinical decision support tools, trainings, technical assistance and quality assurance to support implementation of VA Suicide Risk Identification Strategy. Available to all facilities.
- Audit and Feedback (Experimental): Audit and Feedback will serve as the first stage implementation intervention for sites that do not meet the benchmark for adequate implementation following 9 months of implementation as usual.
  Interventions: Behavioral: Audit and Feedback
- External Facilitation (Experimental): Audit and Feedback plus External Facilitation will serve as the second stage implementation intervention for sites that still do not meet the benchmark for adequate implementation following 9 months of implementation as usual plus audit and feedback.
  Interventions: Behavioral: Audit and Feedback; Behavioral: External Facilitation

INTERVENTIONS:
Behavioral: Audit and Feedback — The following components will be incorporated into the audit and feedback intervention: i) individualized facility performance data (site level), ii) frequent delivery intervals (monthly), iii) comparisons with other sites, iv) graphical and text form displays of information, v) constructive, non-punitive tone, vi) target performance or benchmark provided, and vii) specific actions or recommendations for meeting the target.
  Arms: Audit and Feedback; External Facilitation
Behavioral: External Facilitation — Facilitation will be conducted by a team of facilitators who will employ the facilitation process to improve uptake of VA Risk ID. Trained external facilitators will flexibly deliver the facilitation process utilizing an integrated set of implementation strategies (e.g., stakeholder engagement, identification of barriers and facilitators, education, problem solving, the use of formative data, communication, and ongoing support).
  Arms: External Facilitation

SUMMARY:
The overall objective of this national quality improvement project is to develop an adaptive implementation strategy to improve the implementation of suicide risk screening and evaluation in Veterans Health Administration ambulatory care settings (i.e., VA Risk ID).

DETAILED DESCRIPTION:
VA Risk ID is the largest implementation of population-based suicide risk screening and evaluation in any United States healthcare system to date. Given the considerable scope of this initiative, several strategies have been employed to support national implementation. To facilitate continuous quality improvement, ongoing evaluation of VA Risk ID and interventions to improve implementation of the three-stage screening and evaluation process are needed. This project is intended to help VHA facilities address challenges to implementing VA Risk ID to fidelity using a sequence of evidence-based implementation strategies (audit and feedback followed by audit and feedback plus external facilitation). By doing so, it will ensure that more Veterans are screened and evaluated for suicide risk, which is the basis of effective, patient-centered suicide risk management. By adapting the implementation intervention "dose" based on facility performance and monitoring implementation over time, this project will allow the program office to focus resources where and when needed the most.

ELIGIBILITY:
Inclusion Criteria:

* Intervention occurs at the site/facility level. Up to 140 VHA facilities across the country will participate in the project. Sites will be allocated to various interventions based on performance (i.e., pre-determined benchmarks for adequate implementation).

Exclusion Criteria:

* This is a national quality improvement project. Sites that are randomized to different intervention arms based on performance may refuse to participate in the implementation interventions.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nazanin H. Bahraini, PhD, Principal Investigator — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (1):
- Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bahraini NH, Matarazzo BB, Barry CN, Post EP, Forster JE, Dollar KM, Dobscha SK, Brenner LA. Protocol: examining the effectiveness of an adaptive implementation intervention to improve uptake of the VA suicide risk identification strategy: a sequential multiple assignment randomized trial. Implement Sci. 2020 Jul 22;15(1):58. doi: 10.1186/s13012-020-01019-6. PMID 32698812
- See also: Project Description — https://www.queri.research.va.gov/national_partnered_evaluations/suicide_identification.cfm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 138 VHA facilities were recruited and enrolled. Sites were allocated to different implementation strategies based on performance.
Pre-assignment Details: All sites started with implementation as usual during run-in phase.
Units Other Than Participants: Sites/Facilities
Groups:
- Implementation As Usual: This arm included sites that responded to implementation as usual during run-in and continued with implementation as usual throughout the trial period. There were no sites in Arm 1 as none of the facilities implemented adequately after the run-in phase.
- Audit & Feedback Responders Continue: This arm included sites that did not implement adequately after the run-in phase, received audit & feedback (A&F) in Phase 1, responded to A&F, and continued A&F in Phase 2.
- Audit & Feedback Responders Switch: This arm included sites that did not implement adequately after the run-in phase, received A&F in Phase 1, responded to A&F and switched to A&F Light in Phase 2. (Note. IAU became A&F Light during Phase 2).
- Audit & Feedback Non-Responders Continue: This arm included sites that did not implement adequately after the run-in phase, received A&F in Phase 1, did not respond to A&F, and continued A&F in Phase 2.
- Audit & Feedback Non-Responders Add Facilitation: This arm included sites that did not implement adequately after the run-in phase, received A&F in Phase 1, did not respond to A&F, and accepted and received A&F + External Facilitation in Phase 2. (Note. Only included sites that accepted EF).
- Implementation As Usual to Audit & Feedback Light: This arm included sites that did not implement adequately after the run-in phase, continued with IAU in Phase 1, and received A&F Light in Phase 2. (Note. IAU became A&F Light during Phase 2)
Period: Phase 1 Intervention
Arm/Group | Implementation As Usual | Audit & Feedback Responders Continue | Audit & Feedback Responders Switch | Audit & Feedback Non-Responders Continue | Audit & Feedback Non-Responders Add Facilitation | Implementation As Usual to Audit & Feedback Light
Started | NA; 0 Sites/Facilities (unit of analysis is site/facility level- no individual participants enrolled) | NA; 6 Sites/Facilities (unit of analysis is site/facility level- no individual participants enrolled) | NA; 6 Sites/Facilities (unit of analysis is site/facility level- no individual participants enrolled) | NA; 40 Sites/Facilities (unit of analysis is site/facility level- no individual participants enrolled) | NA; 17 Sites/Facilities (unit of analysis is site/facility level- no individual participants enrolled) | NA; 69 Sites/Facilities (unit of analysis is site/facility level- no individual participants enrolled)
Completed | NA; 0 Sites/Facilities (This arm included sites that responded to implementation as usual during run-in and continued with implementation as usual throughout the trial period. There were no sites in this arm as none of the facilities implemented adequately after the run-in phase. unit of analysis is site/facility level- no individual participants enrolled) | NA; 6 Sites/Facilities (A total of 12 sites responded to audit & feedback during Phase 1. Six sites were randomized to continue audit & feedback during phase 2 and another 6 were randomized to switch to audit & feedback light during phase 2. unit of analysis is site/facility level- no individual participants enrolled) | NA; 6 Sites/Facilities (A total of 12 sites responded to audit & feedback during Phase 1. Six sites were randomized to continue audit & feedback during phase 2 and another 6 were randomized to switch to audit & feedback light during phase 2. unit of analysis is site/facility level- no individual participants enrolled) | NA; 40 Sites/Facilities (29 of the 57 sites that did not respond to audit & feedback during Phase 1, were randomized to continue audit & feedback in phase 2. An additional 11 sites that were randomized to receive external facilitation declined and remained in this group for a total of 40 sites. unit of analysis is site/facility level- no individual participants enrolled) | NA; 17 Sites/Facilities (28 of the 57 sites that did not respond to audit & feedback during Phase 1, were randomized to continue audit & feedback with the addition of external facilitation. 17 sites accepted external facilitation and 11 sites declined. The 11 sites that declined remained in the audit & feedback no response continue group. unit of analysis is site/facility level- no individual participants enrolled) | NA; 69 Sites/Facilities (unit of analysis is site/facility level- no individual participants enrolled)
Not Completed | NA; 0 Sites/Facilities | NA; 0 Sites/Facilities | NA; 0 Sites/Facilities | NA; 0 Sites/Facilities | NA; 0 Sites/Facilities | NA; 0 Sites/Facilities
Period: Phase 2 Intervention
Arm/Group | Implementation As Usual | Audit & Feedback Responders Continue | Audit & Feedback Responders Switch | Audit & Feedback Non-Responders Continue | Audit & Feedback Non-Responders Add Facilitation | Implementation As Usual to Audit & Feedback Light
Started | NA; 0 Sites/Facilities (Unit of analysis is site/facility- no individual participants enrolled) | NA; 6 Sites/Facilities (Unit of analysis is site/facility- no individual participants enrolled) | NA; 6 Sites/Facilities (Unit of analysis is site/facility- no individual participants enrolled) | NA; 40 Sites/Facilities (Unit of analysis is site/facility- no individual participants enrolled) | NA; 17 Sites/Facilities (Unit of analysis is site/facility- no individual participants enrolled) | NA; 69 Sites/Facilities (Unit of analysis is site/facility- no individual participants enrolled)
Completed | NA; 0 Sites/Facilities (Unit of analysis is site/facility- no individual participants enrolled) | NA; 6 Sites/Facilities (Unit of analysis is site/facility- no individual participants enrolled) | NA; 6 Sites/Facilities (Unit of analysis is site/facility- no individual participants enrolled) | NA; 38 Sites/Facilities (Unit of analysis is site/facility- no individual participants enrolled) | NA; 17 Sites/Facilities (The 17 sites represented here reflect sites that accepted EF; all others opted to forgo external facilitation and continue with audit & feedback only. Unit of analysis is site/facility- no individual participants enrolled) | NA; 66 Sites/Facilities (Unit of analysis is site/facility- no individual participants enrolled)
Not Completed | NA; 0 Sites/Facilities | NA; 0 Sites/Facilities | NA; 0 Sites/Facilities | NA; 2 Sites/Facilities | NA; 0 Sites/Facilities | NA; 3 Sites/Facilities

BASELINE CHARACTERISTICS:
Population: Participants are not the unit of analysis; sites/medical centers are the unit of analysis.
Units Other Than Participants: Site/Facilities
Groups:
- Implementation As Usual: This group included sites that responded to implementation as usual during run-in and continued with implementation as usual throughout the trial period. There were no sites in Arm 1 as none of the facilities implemented adequately after the run-in phase.
- Audit & Feedback Responders Continue: This group included sites that did not implement adequately after the run-in phase, received audit & feedback (A&F) in Phase 1, responded to A&F, and continued A&F in Phase 2.
  Phase 1: randomized to A&F arm
  Phase 2: randomized A&F arm again
- Audit & Feedback Responders Switch: This group included sites that did not implement adequately after the run-in phase, received A&F in Phase 1, responded to A&F and switched to A&F Light in Phase 2. (Note. IAU became A&F Light during Phase 2).
  Phase 1: randomized to A&F arm
  Phase 2: randomized A&F Light arm
- Audit & Feedback Non-Responders Continue: This group included sites that did not implement adequately after the run-in phase, received A&F in Phase 1, did not respond to A&F, and continued A&F in Phase 2.
  Phase 1: randomized to A&F arm
  Phase 2: randomized A&F arm again
- Audit & Feedback Non-Responders Add Facilitation: This group included sites that did not implement adequately after the run-in phase, received A&F in Phase 1, did not respond to A&F, and accepted and received A&F + External Facilitation in Phase 2. (Note. Only included sites that accepted EF).
  Phase 1: randomized to A&F arm
  Phase 2: randomized to A&F plus External Facilitation arm
- Implementation As Usual to Audit & Feedback Light: This group included sites that did not implement adequately after the run-in phase, continued with IAU in Phase 1, and received A&F Light in Phase 2. (Note. IAU became A&F Light during Phase 2)
  Phase 1: randomized to Implementation as Usual arm
  Phase 2: received implementation as usual which became A&F Light
- Total: Total of all reporting groups
Arm/Group | Implementation As Usual | Audit & Feedback Responders Continue | Audit & Feedback Responders Switch | Audit & Feedback Non-Responders Continue | Audit & Feedback Non-Responders Add Facilitation | Implementation As Usual to Audit & Feedback Light | Total
Number analyzed (Participants) | NA | NA | NA | NA | NA | NA | NA
Number analyzed (Site/Facilities) | 0 | 6 | 6 | 38 | 17 | 66 | 133
Age, Continuous [Mean (Standard Deviation); unit: years] |  | NA (NA) — unit of analysis is sites; no participants enrolled | NA (NA) — unit of analysis is sites; no participants enrolled | NA (NA) — unit of analysis is sites; no participants enrolled | NA (NA) — unit of analysis is sites; no participants enrolled | NA (NA) — unit of analysis is sites; no participants enrolled | NA (NA) — unit of analysis is sites; no participants enrolled
Sex: Female, Male [Count of Units; unit: Site/Facilities]
  Female |  | NA — unit of analysis is sites; no participants enrolled | NA — unit of analysis is sites; no participants enrolled | NA — unit of analysis is sites; no participants enrolled | NA — unit of analysis is sites; no participants enrolled | NA — unit of analysis is sites; no participants enrolled | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male |  | NA — unit of analysis is sites; no participants enrolled | NA — unit of analysis is sites; no participants enrolled | NA — unit of analysis is sites; no participants enrolled | NA — unit of analysis is sites; no participants enrolled | NA — unit of analysis is sites; no participants enrolled | NA — Total not calculated because data are not available (NA) in one or more arms.
Race (NIH/OMB) [Count of Units; unit: Site/Facilities]
  American Indian or Alaska Native |  | NA — unit of analysis is sites; no participants enrolled | NA — unit of analysis is sites; no participants enrolled | NA — unit of analysis is sites; no participants enrolled | NA — unit of analysis is sites; no participants enrolled | NA — unit of analysis is sites; no participants enrolled | NA — Total not calculated because data are not available (NA) in one or more arms.
  Asian |  | NA — unit of analysis is sites; no participants enrolled | NA — unit of analysis is sites; no participants enrolled | NA — unit of analysis is sites; no participants enrolled | NA — unit of analysis is sites; no participants enrolled | NA — unit of analysis is sites; no participants enrolled | NA — Total not calculated because data are not available (NA) in one or more arms.
  Native Hawaiian or Other Pacific Islander |  | NA — unit of analysis is sites; no participants enrolled | NA — unit of analysis is sites; no participants enrolled | NA — unit of analysis is sites; no participants enrolled | NA — unit of analysis is sites; no participants enrolled | NA — unit of analysis is sites; no participants enrolled | NA — Total not calculated because data are not available (NA) in one or more arms.
  Black or African American |  | NA — unit of analysis is sites; no participants enrolled | NA — unit of analysis is sites; no participants enrolled | NA — unit of analysis is sites; no participants enrolled | NA — unit of analysis is sites; no participants enrolled | NA — unit of analysis is sites; no participants enrolled | NA — Total not calculated because data are not available (NA) in one or more arms.
  White |  | NA — unit of analysis is sites; no participants enrolled | NA — unit of analysis is sites; no participants enrolled | NA — unit of analysis is sites; no participants enrolled | NA — unit of analysis is sites; no participants enrolled | NA — unit of analysis is sites; no participants enrolled | NA — Total not calculated because data are not available (NA) in one or more arms.
  More than one race |  | NA — unit of analysis is sites; no participants enrolled | NA — unit of analysis is sites; no participants enrolled | NA — unit of analysis is sites; no participants enrolled | NA — unit of analysis is sites; no participants enrolled | NA — unit of analysis is sites; no participants enrolled | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported |  | NA — unit of analysis is sites; no participants enrolled | NA — unit of analysis is sites; no participants enrolled | NA — unit of analysis is sites; no participants enrolled | NA — unit of analysis is sites; no participants enrolled | NA — unit of analysis is sites; no participants enrolled | NA — Total not calculated because data are not available (NA) in one or more arms.
Region of Enrollment [Number; unit: Site/Facilities]
  United States |  | 6 | 6 | 38 | 17 | 66 | 133
Facility Complexity [Count of Units; unit: Site/Facilities] — The Facility Complexity Model classifies VA medical facility complexity level based on patient population, clinical services offered, educational and research missions, and administrative complexity. Level-1a facilities are the most complex and level-3 facilities are the least complex. Levels 1a-1c will be considered high complexity, level 2- medium complexity and level 3- low complexity.
  Site/Facilities
    Facility Complexity Level 1a-1c |  | 2 | 1 | 26 | 13 | 41 | 83
    Facility Complexity Level 2 |  | 1 | 1 | 4 | 4 | 12 | 22
    Facility Complexity Level 3 |  | 3 | 4 | 8 | 0 | 13 | 28

OUTCOME MEASURES:

1. Primary Outcome: Change in Columbia Suicide Severity Rating Scale Screener (C-SSRS) Uptake- Phase 1
Description: C-SSRS uptake is a site level adherence measure of the percentage of patients in ambulatory care who received a timely annual suicide risk screen (i.e., during the first encounter/visit after the annual suicide risk screen reminder was due). Adherence ranges from 0 to 100, higher scores reflect higher adherence. The outcome measure is reported as the change in facility adherence from baseline to month 8 of intervention Phase 1. Higher numbers reflect greater change in adherence from baseline to month 8 of intervention Phase 1.
Time Frame: Change from baseline and intervention Phase 1 month 8
Population: All sites that completed Phase 1 are included in the analysis. Sites that received Audit & Feedback in addition to Implementation as Usual during Phase 1 are compared to sites that only received Implementation as Usual during Phase 1.
Measure: Mean (95% Confidence Interval); unit: change in percent adherence
Units Other Than Participants: Sites/Facilities
Groups:
- Phase 1: Audit & Feedback: This arm included sites that received audit and feedback in additional to implementation as usual during Phase 1.
- Phase 1: Implementation As Usual: This arm included all sites that received implementation as usual during Phase 1.
Arm/Group | Phase 1: Audit & Feedback | Phase 1: Implementation As Usual
Number analyzed (Participants) | NA | NA
Number analyzed (Sites/Facilities) | 67 | 66
change in percent adherence | 13.0 [11.9 to 14.0] | 11.9 [10.9 to 13.0]
Statistical Analysis 1: Comparison: Phase 1: Audit & Feedback vs Phase 1: Implementation As Usual; Test type: Superiority; p = 0.18, Mixed Models Analysis — the p-values are not adjusted for multiple comparisons and the a priori threshold for statistical significance is 0.05; Mean Difference (Net) = 1.01, 95% CI 2-sided [-0.46 to 2.48]

2. Primary Outcome: Change in Comprehensive Suicide Risk Evaluation (CSRE) Uptake- Phase 1
Description: CSRE uptake is a site level adherence measure of the percentage of patients in ambulatory care who had a positive C-SSRS screener and received the CSRE as intended (same day and by the appropriate provider). The score is a facility adherence score. Adherence ranges from 0 to 100, higher scores reflect higher adherence. The outcome measure is reported as the change in facility adherence from baseline to month 8 of intervention Phase 1. Higher numbers reflect greater change in adherence from baseline to month 8 of intervention Phase 1.
Time Frame: Change from baseline and intervention Phase 1 month 8
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: change in percent adherence
Units Other Than Participants: Sites/Facilities
Groups:
- Phase 1: Audit & Feedback: This arm includes all sites that received audit & feedback in addition to implementation as usual during Phase 1.
Arm/Group | Phase 1: Audit & Feedback | Phase 1: Implementation As Usual
Number analyzed (Participants) | NA | NA
Number analyzed (Sites/Facilities) | 67 | 66
change in percent adherence | 11.0 [8.43 to 13.6] | 7.45 [4.82 to 10.1]
Statistical Analysis 1: Comparison: Phase 1: Audit & Feedback vs Phase 1: Implementation As Usual; Test type: Superiority; p = .06, Mixed Models Analysis — the p-values are not adjusted for multiple comparisons and the a priori threshold for statistical significance is 0.05; Mean Difference (Net) = 3.58, 95% CI 2-sided [-0.11 to 7.28]

3. Secondary Outcome: Change in Columbia Suicide Severity Rating Scale Screener (C-SSRS) Uptake- Phase 2a
Description: C-SSRS uptake is a site level adherence measure of the percentage of patients in ambulatory care who received a timely annual suicide risk screen (i.e., during the first encounter/visit after the annual suicide risk screen reminder was due). The score is a facility adherence score. Adherence ranges from 0 to 100, higher scores reflect higher adherence. The outcome measure is reported as the change in facility adherence from month 9 of intervention phase 1 to month 9 of intervention phase 2. Higher numbers reflect greater change in adherence from month 9 of intervention phase 1 to month 9 of intervention phase 2.
Time Frame: Change from month 9 of intervention phase 1 and month 9 of intervention phase 2
Population: Responding sites that continued to received audit & feedback during Phase 2 are compared to responding sites that switched to audit & feedback light during Phase 2. For Phase 2, it was pre-specified to compare only Audit & Feedback Light to Audit and Feedback for the group of sites that responded to Audit & Feedback during Phase 1.
Measure: Mean (95% Confidence Interval); unit: change in percent adherence
Units Other Than Participants: Sites/Facilities
Groups:
- Phase 2a: Responders Audit & Feedback: This arm includes sites that responded to audit & feedback during Phase 1 and continued to receive audit & feedback during Phase 2.
- Phase 2a: Responders Audit & Feedback Light: This arm included sites that responded to audit and feedback during Phase 1 and were switched to Audit & Feedback Light during Phase 2.
Arm/Group | Phase 2a: Responders Audit & Feedback | Phase 2a: Responders Audit & Feedback Light
Number analyzed (Participants) | NA | NA
Number analyzed (Sites/Facilities) | 6 | 6
change in percent adherence | 13.3 [9.0 to 17.7] | 11.7 [7.3 to 16.0]
Statistical Analysis 1: Comparison: Phase 2a: Responders Audit & Feedback vs Phase 2a: Responders Audit & Feedback Light; Test type: Superiority; p = 0.60, Mixed Models Analysis — the p-values are not adjusted for multiple comparisons and the a priori threshold for statistical significance is 0.05; Median Difference (Net) = 1.7, 95% CI 2-sided [-4.5 to 7.9]

4. Secondary Outcome: Change in Comprehensive Suicide Risk Evaluation (CSRE) Uptake-Phase 2a
Description: CSRE uptake is a site level adherence measure of the percentage of patients in ambulatory care who had a positive C-SSRS screener and received the CSRE as intended (same day and by the appropriate provider). The score is a facility adherence score. Adherence ranges from 0 to 100, higher scores reflect higher adherence. The outcome measure is reported as the change in facility adherence from month 9 of intervention phase 1 to month 9 of intervention phase 2. Higher numbers reflect greater change in adherence from month 9 of intervention phase 1 to month 9 of intervention phase 2.
Time Frame: Change from month 9 of intervention phase 1 and month 9 of intervention phase 2
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: change in percent adherence
Units Other Than Participants: Sites/Facilities
Arm/Group | Phase 2a: Responders Audit & Feedback | Phase 2a: Responders Audit & Feedback Light
Number analyzed (Participants) | NA | NA
Number analyzed (Sites/Facilities) | 6 | 6
change in percent adherence | 6.2 [0.02 to 12.3] | 10.2 [4.0 to 16.5]
Statistical Analysis 1: Comparison: Phase 2a: Responders Audit & Feedback vs Phase 2a: Responders Audit & Feedback Light; Test type: Superiority; p = 0.36, Mixed Models Analysis — p-values are not adjusted for multiple comparisons and the a priori threshold for statistical significance is 0.05; Median Difference (Net) = -4.1, 95% CI 2-sided [-12.8 to 4.7]

5. Secondary Outcome: Change in Columbia Suicide Severity Rating Scale Screener (C-SSRS) Uptake- Phase 2b
Description: as for outcome 3
Time Frame: Change from month 9 of intervention phase 1 and month 9 of intervention phase 2
Population: Nonresponding sites that received audit and feedback in Phase 2 are compared to nonresponding sites that received audit & feedback plus external facilitation during Phase 2.
Measure: Mean (95% Confidence Interval); unit: change in percent adherence
Units Other Than Participants: Sites/Facilities
Groups:
- Phase 2b: Nonresponders Audit & Feedback: This arm included sites that did not respond to audit & feedback during Phase 1 and continued to received audit & feedback during Phase 2.
- Phase 2b: Nonresponders External Facilitation: This arm included sites that did not respond to Audit & Feedback during Phase 1 and received External Facilitation in addition to Audit & Feedback during Phase 2. (Note. Only included sites that accepted external facilitation).
Arm/Group | Phase 2b: Nonresponders Audit & Feedback | Phase 2b: Nonresponders External Facilitation
Number analyzed (Participants) | NA | NA
Number analyzed (Sites/Facilities) | 38 | 17
change in percent adherence | 18.9 [16.8 to 21.0] | 23.4 [20.2 to 26.5]
Statistical Analysis 1: Comparison: Phase 2b: Nonresponders Audit & Feedback vs Phase 2b: Nonresponders External Facilitation; Test type: Superiority; p = .02, Mixed Models Analysis — p-values are not adjusted for multiple comparisons and the a priori threshold for statistical significance is 0.05; Mean Difference (Net) = -4.5, 95% CI 2-sided [-8.3 to -0.67]

6. Secondary Outcome: Change in Comprehensive Suicide Risk Evaluation (CSRE) Uptake-Phase 2b
Description: as for outcome 4
Time Frame: Change from month 9 of intervention phase 1 and month 9 of intervention phase 2
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: change in percent adherence
Units Other Than Participants: Sites/Facilities
Arm/Group | Phase 2b: Nonresponders Audit & Feedback | Phase 2b: Nonresponders External Facilitation
Number analyzed (Participants) | NA | NA
Number analyzed (Sites/Facilities) | 38 | 17
change in percent adherence | 13.0 [10.3 to 15.7] | 13.6 [9.5 to 17.7]
Statistical Analysis 1: Comparison: Phase 2b: Nonresponders Audit & Feedback vs Phase 2b: Nonresponders External Facilitation; Test type: Superiority; p = 0.82, Mixed Models Analysis; Mean Difference (Net) = -0.56, 95% CI 2-sided [-5.5 to 4.4]

ADVERSE EVENTS:
Time Frame: No adverse event data were collected.
Arm/Group | Implementation As Usual | Audit & Feedback Responders Continue | Audit & Feedback Responders Switch | Audit & Feedback Non-Responders Continue | Audit & Feedback Non-Responders Add Facilitation | Implementation As Usual to Audit & Feedback Light
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Shortened study timeline due to COVID; study phases needed to be shortened potentially limiting ability to detect an impact of phase 1 intervention- audit & feedback

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT04243330/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-17): https://cdn.clinicaltrials.gov/large-docs/30/NCT04243330/SAP_001.pdf